CLINICAL TRIAL: NCT04907214
Title: The Effect of SGLT2 Inhibition on Adipose Tissue Inflammation and Endothelial Function Pilot
Brief Title: SGLT2 Inhibitor Effects on Inflammation and Heart Disease in Obesity Pilot
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mona Mashayekhi, Clinical Instructor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 210907
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Pre-diabetes
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental): Individuals receive empagliflozin 25mg/day orally for 12 weeks
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Oral empagliflozin daily

SUMMARY:
Obesity is associated with increased cardiometabolic disease risk due, in part, to heightened chronic inflammation arising from adipose tissue. There are no current targeted therapies to prevent or reverse the chronic inflammation of obesity, and a better understanding of these inflammatory pathways in humans is key to future therapeutic interventions. This project will determine both the anti-inflammatory potential of the SGLT2 inhibitor empagliflozin, and the contribution of adipose inflammation to surrogate measures of cardiovascular disease in a randomized controlled trial of obese patients.

DETAILED DESCRIPTION:
This study will be expanded to include another 10 participants. Enrollment will begin July 1, 2023.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 to 70 years old
2. Impaired glucose tolerance (two-hour plasma glucose 140-199 mg/dL) or impaired fasting glucose (100-125mg/dL) or HbA1c 5.7-6.4%
3. BMI ≥ 30 kg/M2
4. The ability to provide informed consent

Exclusion criteria:

Criteria Related to Medical Diagnoses/Conditions/Treatments:

1. Diabetes type 1 or type 2, as defined by a fasting plasma glucose of 126 mg/dL or greater, a two-hour plasma glucose of 200 mg/dL or greater, HbA1c ≥6.5%, or the use of anti-diabetic medication
2. Pregnancy or breast-feeding. Women of child-bearing potential will be required to have undergone tubal ligation or to be using an oral contraceptive or barrier methods of birth control
3. Cardiovascular disease such as myocardial infarction within six months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
4. Presence of implanted cardiac defibrillator or pacemaker
5. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
6. History of pancreatitis or pancreatic surgery
7. History or presence of immunological or hematological disorders
8. Clinically significant gastrointestinal impairment that could interfere with drug absorption
9. History of advanced liver disease with cirrhosis
10. Individuals with an eGFR<45 mL/min/1.73 m2, where eGFR is determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine is expressed in mg/dL and age in years: eGFR (mL/min/1.73m2)=186 • Scr-1.154 • age-0.203 • (0.742 if female)
11. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
12. Treatment with anticoagulants
13. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
14. History of alcohol abuse (>14 per week for men and >7 per week for women) or illicit drug use
15. Treatment with any investigational drug in the one month preceding the study
16. Previous randomization in this trial
17. Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
18. Inability to comply with the protocol in the opinion of the principal investigator, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

    Criteria Related to Known Adverse Effects of Drug:
19. Uncircumcised men or men with history of balanitis
20. History of urinary incontinence
21. History of recurrent (>3) episodes of vulvovaginitis per year, or severe symptoms
22. History of Fournier's gangrene
23. History of recurrent (≥3) UTIs per year or pyelonephritis
24. History of symptomatic hypotension or conditions predisposing to volume depletion
25. Known peripheral vascular disease, neuropathy, history of foot ulcers or lower limb amputations
26. Treatment with loop diuretics furosemide, torsemide, bumetanide, ethacrynic acid
27. Known or suspected allergy to trial medications, excipients, or related products
28. Contraindications to study medications, worded specifically as stated in the product's prescribing information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mashayekhi, MD/PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * 17 in the Original study + 21 in the Extension study signed consent for a total of 38.
  * 9 individuals in the Extension study did not perform screening procedures after consent and were not enrolled. In total 29 individuals enrolled.
  * 11 individuals in the Original study and 2 individuals in the Extension study did not meet inclusion/exclusion criteria after screening.
  * 6 individuals in the Original study and 10 individuals in the Extension study started and completed study days.
Period: Overall Study
Arm/Group | Empagliflozin
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Empagliflozin
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Pro-inflammatory T helper type 1 cells in adipose tissue [Mean (Standard Deviation); unit: Percentage of CD3+ T cells] — Population: -One individual could not tolerate the liposuction and did not provide a sample.
  Percentage of CD3+ T cells
    number analyzed (Participants) | 5
    (all) | 13.0 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adipose Pro-inflammatory T Helper Type 1 Cell Percentages After 3 Months
Description: Pro-inflammatory T helper type 1 cells are quantified using flow cytometry
Time Frame: Baseline to 12 weeks
Population: One individual did not tolerate the liposuction technique and did not provide adipose tissue for the study.
Measure: Mean (Standard Deviation); unit: Percentage of CD3+ T cells
Arm/Group | Empagliflozin
Number analyzed (Participants) | 5
Percentage of CD3+ T cells | -1.6 (1.8)

2. Primary Outcome: Change in Flow-mediated Dilation After 3 Months
Description: Endothelial function quantified using flow-mediated dilation by ultrasound, measuring percentage increase in artery diameter during hyperemia.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change in diameter
Arm/Group | Empagliflozin
Number analyzed (Participants) | 6
Percentage change in diameter | -2.33 (7.72)

3. Primary Outcome: Change in Liver Steatosis at 3 Months
Description: Liver steatosis assessment by transient elastography-controlled attenuation parameter imaging, reported as Controlled Attenuation Parameter (CAP)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Decibels per meter
Arm/Group | Empagliflozin
Number analyzed (Participants) | 6
Decibels per meter | 0.17 (28.12)

4. Secondary Outcome: Change in Adipose Pro-inflammatory T Helper Type 1 Cell Percentages After 2 Weeks
Description: Pro-inflammatory T cells are quantified using flow cytometry
Time Frame: Baseline to 2 weeks
Population: One individual did not tolerate the liposuction technique and did not provide adipose tissue for the study.
Measure: Mean (Standard Deviation); unit: Percentage of CD3+ T cells
Arm/Group | Empagliflozin
Number analyzed (Participants) | 5
Percentage of CD3+ T cells | -0.5 (5.0)

5. Secondary Outcome: Change in the Plasma Inflammatory Cytokine IL-6 After 3 Months
Description: IL-6 is quantified in plasma samples.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: picogram per milliliter
Arm/Group | Empagliflozin
Number analyzed (Participants) | 6
picogram per milliliter | 0.078 (0.717)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Empagliflozin
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empagliflozin (N=6)
Skin infection (Skin and subcutaneous tissue disorders) | 1 — Bacterial skin infection of tattoo, requiring Bactrim for 10 days.
Headache (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04907214/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04907214/ICF_000.pdf